CLINICAL TRIAL: NCT04311476
Title: Autologous Cord Blood Cells for Prevention of BPD in Preterm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: yangjie (Other)
Responsible Party: Sponsor-Investigator, yangjie, Director of Dept of Neonatology, Guangdong Women and Children Hospital
Organization: Guangdong Women and Children Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Guangdong WC H
Record Dates: First submitted 2020-03-15; First posted 2020-03-17 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Safety Issues; BPD - Bronchopulmonary Dysplasia; Neonatal Death
Keywords: ACBMNC; very premature infants; BPD
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Perinatal Death

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 0.9% sodium chloride infusion within 24 hours after birth
  Interventions: Drug: 0.9% Sodiun Chloride
- ACBMNC (Experimental): Autologous Umbilical Cord Blood Mononuclear Cells intravenously within 24 hours after birth,dose is 5×107cells/kg ,
  Interventions: Other: Autologous Umbilical Cord Blood Mononuclear Cells infusion Therapy

INTERVENTIONS:
Other: Autologous Umbilical Cord Blood Mononuclear Cells infusion Therapy — Evaluate Autologous cord blood cells infusion on prevention of bronchopulmonary dysplasia in very preterm neonates
  Other Names: Autologous Umbilical Cord Blood Mononuclear Cells Therapy
  Arms: ACBMNC
Drug: 0.9% Sodiun Chloride — 0.9% Sodiun Chloride in control group
  Arms: Placebo

SUMMARY:
To study the effect of Autologous cord blood cells infusion on prevention of bronchopulmonary dysplasia in very preterm neonates

DETAILED DESCRIPTION:
We did a randomized, double-blind, placebo-controlled trial to assess effect of one intravenous dose of cord blood MNCs compared with placebo in reducing incidence of BPD in very preterm neonates.We enrolled preterm neonates less than 32 weeks of GA at neonatal intensive care units (NICUs) in Guangdong Women and Children Hospital within the first 24 postnatal hours. Patients were randomly assigned by 1:1 to receive either (5×107cells/kg ACBMNC or normal saline intravenously within 24 hours after birth according to a computer-generated schedule. The primary endpoint was efficacy at 36 GA or discharge home and all analyses were done by intention to prevent.MNCs viability was also tested before transfusion

ELIGIBILITY:
Inclusion Criteria:

* born in the study hospital;
* singleton birth;
* less than 32 weeks GA
* Without congenital malformations or known chromosomal aberrations;
* Without clinical chorioamnionitis;
* the mother was negative for hepatitis B (HBsAg and/or HBeAg) and C virus (anti-HCV), syphilis, HIV (anti-HIV-1 and -2) and IgM against cytomegalovirus, rubella, toxoplasma and herpes simplex virus;
* consents were obtained from their parents or guardians;
* the umbilical cord blood cells after processing were available.

Exclusion Criteria:

* birth-weight was less than the third percentile for gestational age according to Fenton curve,
* if they had severe perinatal asphyxia (defined as an Apgarscore of 0-3 for more than 5 minutes, a cord blood pH of less than 7.00, or both) and were expected to die shortly after birth.

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
number of patients without bronchopulmonary dysplasia | at 36 weeks of postmenstrual age or discharge home, whichever came first
  bronchopulmonary dysplasia incidence

SECONDARY OUTCOMES:
number of patients who died， severe bronchopulmonary dysplasia | at 36 weeks of postmenstrual age
  mortaliity rate

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, PHD, Principal Investigator — Guangdong Women and Children Hospital
Locations (1):
- Jie Yang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No